CLINICAL TRIAL: NCT01205100
Title: Feedback-assisted Treatment of Abdominal Distension - a Randomized Controlled Trial
Brief Title: Treatment of Abdominal Distension by Biofeedback - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)60/2009
Record Dates: First submitted 2010-09-06; First posted 2010-09-20 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia
Keywords: Gastrointestinal Diseases; Irritable Bowel Syndrome; Behavioral Research; Biofeedback
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback (Active Comparator): Patients will be taught to control abdominal and diaphragmatic muscles by bio-feedback using EMG recordings.
  Interventions: Behavioral: Bio-feedback
- Placebo medication (Placebo Comparator): Electromyography will be recorded but not shown to the patients. Patients will take a pill of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Bio-feedback — By providing on-line electromyography information of muscle activity, patients will be able to control and actively correct their muscle activity during the 15 min treatment session. Each patients will attend 3 treatment sessions.
  Arms: Biofeedback
Drug: Placebo
  Arms: Placebo medication

SUMMARY:
Background: Abdominal bloating is a frequent and bothersome complaint in patients with functional gut disorders without satisfactory treatment to date. Recent data from our laboratory indicate that abdominal distention in these patients is produced by abdomino-phrenic dyssynergia: diaphragmatic contraction associated with abdominal wall relaxation (particularly the internal oblique). In analogy to other clinical situations (e.g. functional outlet obstruction, rumination or aerophagia) behavioral treatment by means of biofeedback might be equally effective in these patients. The investigators hypothesized that abdomino-phrenic coordination and abdominal distention can be controlled by biofeedback techniques.

Aim: to prove the efficacy of behavioural treatment using biofeedback techniques for abdominal distension.

Randomization: Patients will be randomized into biofeedback and placebo groups.

Intervention. Biofeedback: patients will be taught to control abdominothoracic muscular activity by bio-feedback using online electromyography information. Placebo: patients will be given a pill containing placebo medication. Interventions will be delivered in 3 sessions (20 min each) over 10-day period

. Measurements: Sensation of abdominal distension will be assessed by means of graphic rating scales graded from 0 (no perception) to 6 (very intense sensation). The activity of the abdomino-thoracic muscles will be recorded. Abdominal distension will be measured by a metric tape fixed to a non-stretch belt placed over the umbilicus.

Outcomes: Primary outcome: Change in sensation of abdominal sensation. Secondary outcomes: a) changes in thoraco-abdominal activity of the muscular walls; activity of thoraco-abdominal muscles (intercostals, diaphragm, external oblique, internal oblique, upper rectus, lower rectus) will be measured by electromyography; b) changes in girth; abdominal girth will be measured using a nonstretch belt (48mm wide) that is placed over the umbilicus. The overlapping ends of the belt will be adjusted carefully with two elastic bands to adapt constantly to the abdominal wall.

ELIGIBILITY:
Inclusion Criteria: episodes of visible abdominal distension triggered by meal ingestion

Exclusion Criteria: organic cause detected by clinical work-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensation of abdominal distension | 10 days
  Sensation score measured by 0-6 scales after each meal (breakfast, lunch, dinner) over a 10-day clinical evaluation period before and after intervention.

SECONDARY OUTCOMES:
Changes in thoraco-abdominal activity of the muscular walls. | 10 days
  Activity of thoraco-abdominal muscles (intercostals, diaphragm, external oblique, internal oblique, upper rectus, lower rectus) will be continuously measured by electromyography.
Changes in girth | 10 days
  Abdominal girth will be continuously measured using a nonstretch belt (48mm wide) that is placed over the umbilicus and ﬁxed to the skin on the back to prevent slipping. The overlapping ends of the belt will be adjusted carefully with two elastic bands to adapt constantly to the abdominal wall. Measurements will be taken before and at the beginning at the end of each intervention session.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, M.D., Principal Investigator — University Hospital Vall d'Hebron
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication in scientific journal.

REFERENCES:
- [Background] Tremolaterra F, Villoria A, Azpiroz F, Serra J, Aguade S, Malagelada JR. Impaired viscerosomatic reflexes and abdominal-wall dystony associated with bloating. Gastroenterology. 2006 Apr;130(4):1062-8. doi: 10.1053/j.gastro.2005.12.036. PMID 16618400
- [Background] Villoria A, Azpiroz F, Soldevilla A, Perez F, Malagelada JR. Abdominal accommodation: a coordinated adaptation of the abdominal wall to its content. Am J Gastroenterol. 2008 Nov;103(11):2807-15. doi: 10.1111/j.1572-0241.2008.02141.x. Epub 2008 Sep 10. PMID 18786126
- [Derived] Barba E, Accarino A, Azpiroz F. Correction of Abdominal Distention by Biofeedback-Guided Control of Abdominothoracic Muscular Activity in a Randomized, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1922-1929. doi: 10.1016/j.cgh.2017.06.052. Epub 2017 Jul 11. PMID 28705783